CLINICAL TRIAL: NCT00526786
Title: A Prospective, Multi-center, Longitudinal Cohort Study of CryoSpray Ablation of Low Grade or High Grade Dysplasia Within Barrett's Esophagus (LCS Dysplasia)
Brief Title: Study of CryoSpray Ablation of Low Grade or High Grade Dysplasia Within Barrett's Esophagus
Acronym: ICE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-00016-00
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Barrett's Esophagus; High Grade Dysplasia; Low Grade Dysplasia
Keywords: Low Grade Dysplasia; High Grade Dysplasia; Barrett's Esophagus; Cryospray ablation; ICE; Cryotherapy; Cryo; CryoSpray
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CryoSpray Ablation System (510(k) NO: K070893) — no drug interventions specified
  Other Names: 510(k) NO: K070893

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the CryoSpray Ablation System to treat esophageal low grade dysplasia (LGD) or high grade dysplasia (HGD) within Barrett's Esophagus (BE).

DETAILED DESCRIPTION:
The study will consist of an estimated 200 subjects with HGD or LGD within BE who are deemed inoperable or refuse standard surgical treatment. A maximum of 20 investigational sites will participate with a maximum of ten subjects per site.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status of 50-100%
* Life expectancy greater than 5 years
* Hematopoietic, Hepatic and Renal lab clearance
* Previous endoscopy with histological confirmation of LGD or HGD within BE
* For Group 2, deemed inoperable based on the following criteria: co-morbid conditions such as severe heart, lung, kidney or liver disease; or refusal of surgical intervention after a thorough unbiased discussion of surgery.
* For Group 2, endoscopic ultrasound (EUS) evaluation demonstrating no evidence of invasion or metastatic lymph node involvement (T0N0M0 by EUS).

Exclusion Criteria:

* Pregnant, not practicing adequate contraception, intending to become pregnant, or lactating at any time during the study (approximately 2 years).
* Esophageal stricture preventing passage of endoscope or catheter.
* Active esophagitis
* EMR performed less than 8 weeks prior to CSA treatment.
* EMR performed on greater than 90% circumference of any area of the esophagus.
* Any previous esophageal surgery, except fundoplication without complications.
* Known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines.
* Concurrent enrollment in an investigational drug or device trial that clinically interferes with the LCS Dysplasia endpoints.
* Psychiatric or other illness deemed by the investigator as an inability to comply with this protocol.
* Medically unfit or other contraindication to tolerate upper endoscopy.
* Inability to tolerate therapy with a proton pump inhibitor (PPI).
* Refusal or inability to give consent.
* Other active malignancy (except nonmelanoma skin cancer or another cancer for which patient is deemed disease-free).
* Concurrent chemotherapy.
* Prior radiation therapy which involved the esophagus.
* Prior adenocarcinoma involving the esophagus or stomach.
* Prior or concurrent ablation therapy including, but not limited to, photodynamic therapy, multipolar electro coagulation, argon plasma coagulation, laser treatment, radio frequency, etc.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The eradication of LGD and HGD within BE at 24 months after the final treatment. The primary safety endpoint is the incidence of all adverse events. | 2 years post treatment

SECONDARY OUTCOMES:
1.Eradication of all BE by 24 months after the final treatment. 2.The proportion of lesions that decreased in length by the 24-month follow-up. 3.The proportion of lesions where severity was downgraded by the 24-month follow-up. | 2 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Greenwald, M.D., Principal Investigator — University of Maryland
Locations (16):
- United States (16):
  - University of California -Irvine, Orange, California
  - Norwalk Hospital, Norwalk, Connecticut
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hoboken Universtiy Medical Center, Hoboken, New Jersey
  - Columbia University Medical Center, New York, New York
  - Universtiy of North Carloina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Lancaster Reginal Medical Center, Lancaster, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Baylor University, Dallas, Texas

REFERENCES:
- [Background] Champion G, Richter JE, Vaezi MF, Singh S, Alexander R. Duodenogastroesophageal reflux: relationship to pH and importance in Barrett's esophagus. Gastroenterology. 1994 Sep;107(3):747-54. doi: 10.1016/0016-5085(94)90123-6. PMID 8076761
- [Background] Eisen GM, Sandler RS, Murray S, Gottfried M. The relationship between gastroesophageal reflux disease and its complications with Barrett's esophagus. Am J Gastroenterol. 1997 Jan;92(1):27-31. PMID 8995932
- [Background] Ell C, May A, Gossner L, Pech O, Gunter E, Mayer G, Henrich R, Vieth M, Muller H, Seitz G, Stolte M. Endoscopic mucosal resection of early cancer and high-grade dysplasia in Barrett's esophagus. Gastroenterology. 2000 Apr;118(4):670-7. doi: 10.1016/s0016-5085(00)70136-3. PMID 10734018
- [Background] Johnston CM, Schoenfeld LP, Mysore JV, Dubois A. Endoscopic spray cryotherapy: a new technique for mucosal ablation in the esophagus. Gastrointest Endosc. 1999 Jul;50(1):86-92. doi: 10.1016/s0016-5107(99)70352-4. PMID 10385730
- [Background] Johnston MH. Cryotherapy and other newer techniques. Gastrointest Endosc Clin N Am. 2003 Jul;13(3):491-504. doi: 10.1016/s1052-5157(03)00044-8. PMID 14629105
- [Background] Johnston MH, Eastone JA, Horwhat JD, Cartledge J, Mathews JS, Foggy JR. Cryoablation of Barrett's esophagus: a pilot study. Gastrointest Endosc. 2005 Dec;62(6):842-8. doi: 10.1016/j.gie.2005.05.008. PMID 16301023